CLINICAL TRIAL: NCT05204407
Title: Luteolin for the Treatment of People With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of California, Los Angeles (Other); Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Robert Buchanan, Chief, Maryland Psychiatric Research Center, Outpatient Research Program, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00099288
Record Dates: First submitted 2022-01-11; First posted 2022-01-24 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Luteolin

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, parallel group, randomized clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Luteolin (Active Comparator)
  Interventions: Dietary Supplement: Luteolin
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Luteolin — The luteolin target dose will be 300 mg BID taken over 12 weeks in capsule form
  Other Names: PureLut
  Arms: Luteolin
Dietary Supplement: Placebo — The placebo target dose will be 300 mg BID taken over 12 weeks in capsule form
  Arms: Placebo

SUMMARY:
Luteolin is a natural product found in foods such as celery, green pepper, parsley, and chamomile tea. It has been found to have anti-cancer, anti-oxidant, and anti-inflammatory properties. The purpose of this study is to determine if luteolin helps improve symptoms of schizophrenia.

DETAILED DESCRIPTION:
The study is a 12-week, double-blind, placebo-controlled, parallel group, randomized clinical trial of the efficacy of luteolin for the treatment of people with schizophrenia, who present with residual symptoms and cognitive impairments. The study will be conducted at two sites: The Maryland Psychiatric Research Center (MPRC) and the University of California Los Angeles (UCLA). Participants will be randomized to either 300mg BID luteolin (three 100mg capsules) or placebo. We hypothesize that luteolin will have significant beneficial effects on global psychopathology and cognitive impairments; decrease antioxidant stress and levels of inflammatory markers; and that improvement in global psychopathology and cognition will be associated with changes in the oxidative stress and inflammatory measures. We also hypothesize that luteolin will be associated with improvements in positive and negative symptoms of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Either male or female of any race
* Age is 18-60 years old
* Meets DSM-5 criteria for schizophrenia or schizoaffective disorder
* Positive and Negative Syndrome Scale (PANSS) total score of 75 or more OR a Clinical Global Impression severity of illness item score of 4 or more
* Clinically stable
* Treated with the same antipsychotic for at least 60 days and have received a constant therapeutic dose for at least 30 days prior to study entry
* Able to participate in the informed consent process and provide voluntary informed consent

Exclusion Criteria:

* Meets DSM-5 criteria for alcohol or substance misuse (except caffeine and nicotine) within the last 6 months; or a positive baseline urine drug screen. Participants who meet DSM-5 criteria for marijuana misuse - mild will be included in the study
* A current infection, including HIV and Hepatitis C; or an organic brain disorder or medical condition, whose pathology or treatment could alter the presentation or treatment of schizophrenia or significantly increase the risk associated with the proposed treatment protocol
* Currently taking immunosuppressive medications (e.g. oral scheduled corticosteroids, chemotherapy or transplantation or HIV/AIDs associated drugs); or anti-inflammatory medications, including NSAIDs (e.g. ibuprofen, celecoxib, or naproxen) or aspirin > 81 mg on a daily basis. The use of PRN anti-inflammatory agents will be allowed.
* Female participants who are pregnant or nursing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2026-01-14 (Actual); Study Completion 2026-01-14 (Actual)

PRIMARY OUTCOMES:
Global psychopathology | 12 weeks
  To determine if luteolin is superior to placebo for the treatment of global psychopathology.
Cognitive impairments | 12 weeks
  To determine if luteolin is superior to placebo for the treatment of cognitive impairments.
Global oxidative stress | 12 weeks
  To determine if luteolin compared to placebo is associated with a decrease in the global measure of oxidative stress and/or a reduction in the levels of the inflammatory markers.
Cognition and oxidative stress | 12 weeks
  To determine if changes in symptom or cognitive measures are associated with changes in the global measure of oxidative stress and/or the levels of inflammatory markers

SECONDARY OUTCOMES:
Positive symptoms of schizophrenia | 12 weeks
  To determine if luteolin is superior to placebo for positive symptoms.
Negative symptoms of schizophrenia | 12 weeks
  To determine if luteolin is superior to placebo for negative symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Buchanan, M.D., Principal Investigator — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - Maryland Psychiatric Research Center, Baltimore, Maryland